CLINICAL TRIAL: NCT02912403
Title: Ambulatory Blood Pressure and the Normal Increase in Maternal Blood Pressure Postpartum
Status: Withdrawn | Type: Observational
Why Stopped: Unable to enroll
Sponsor: St. Louis University (Other)
Responsible Party: Principal Investigator, Jennifer Goldkamp, MD, MD, St. Louis University
Other Study IDs: 27285
Record Dates: First submitted 2016-08-22; First posted 2016-09-23 (Estimated); Last update posted 2017-03-06 (Actual); Status verified 2017-03

CONDITIONS: Normotensive Postpartum Cesarean Section Patients

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Postpartum Cesarean Section: We will be including postpartum women as this study idea is pertaining to recent pregnancy

SUMMARY:
Investigators plan to study blood pressure trends on days 3 to 6 of the postpartum period. Investigators will use a home blood pressure monitor that stays on the arm, and takes blood pressures hourly. Participants will record any symptoms that they feel are attributed to high blood pressure and pain medication use.

DETAILED DESCRIPTION:
Participants will be screened postpartum for inclusion. Only women with cesarean deliveries will be included as they are kept for 3 days in the hospital as opposed to 2 days for vaginal deliveries. If they meet inclusion criteria they will be asked to participate in the study, and consented. Each patient will receive routine postpartum care. The ambulatory blood pressure cuff will be introduced and validated on the particpant prior to discharge. Particpants will then be given specific instructions on when to place the cuff on their am and when to remove it. The ambulatory cuff will take blood pressure measurements every hour. The Particpant will be asked to keep a log of actives, symptoms, and pain medication use for the 72 hour period that her blood pressures are being recorded. The BP device will be returned to the department of OB/GYN at St. Mary's after completion of her 72 hours of monitoring. This will occur at her first post op visit. Particpants will be asked to complete a survey about comfort of device and return with the device. Information pertaining to their pregnancy and delivery will be collected while the patient is in the hospital. Particpants are not responsible for damage or loss of equipment.

All of these procedures are part of the study.

ELIGIBILITY:
Inclusion Criteria:

* Normotensive postpartum women
* Singleton pregnancy
* Cesarean delivery

Exclusion Criteria:

* Chronic medical conditions that would put the patient at increased risk for hypertension (diabetes, lupus, renal disease)
* Current diagnosis of hypertensive disease
* Skin rash in location of cuff placement
* Tobacco user
* Chronic narcotic user
* Vaginal delivery
* cognitively impaired persons

Ages: 14 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: postpartum women
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-08 (Estimated); Primary Completion 2017-08 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
blood pressure changes on days 3 to 6 of the postpartum period | days 3 to 6 of the postpartum period
  To determine the normal blood pressure trends for women with uncomplicated pregnancies during days 3 to 6 of the postpartum period. These days are historically considered the "at risk days" for rising blood pressures.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Goldkamp, MD, Principal Investigator — St. Louis University
Locations (1):
- St. Mary's Health Center, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No